CLINICAL TRIAL: NCT00815737
Title: Effectiveness and Safety of Rhubarb for the Treatment of Patients Who Have Suffered From Cerebral Hemorrhage
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Zhongshan hospital, Fudan University, TCM department, Zhongshan hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rhubarb cerebral hemorrhage
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2009-09

CONDITIONS: Lung Infection; Cerebral Hemorrhage; Pneumonia
Keywords: Lung Infection After Cerebral Hemorrhage; Prevention of Pneumonia; Rhubarb
MeSH Terms: conditions — Cerebral Hemorrhage; Pneumonia | interventions — rhubarb peony decoction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Experimental)
  Interventions: Drug: rhubarb
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rhubarb — 14 days of rhubarb
  Arms: A
Drug: Placebo — 14 days of Placebo
  Arms: B

SUMMARY:
This study will determine if rhubarb will reduced the incidence of pneumonia and improved recovery from an acute cerebral hemorrhage. The study is designed to look at both infection rate and overall recovery and recovery of motor function, for example muscle strength and coordination.

ELIGIBILITY:
Inclusion Criteria:

* Occurrence of an acute cerebral hemorrhage (between 9 and 72 h after onset) with a score of at least 6 on the National Institute of Health Stroke Scale (NIHSS), and patient age of at least 18 years.
* Have no pneumonia according to modified criteria of the U.S. Centers for Disease Control and Prevention (CDC)
* Consistent with the Constipation of Phlegm-Heat Accumulation type by Traditional Chinese Medicine (TCM) standard
* Patients or their representatives voluntarily take part in this study and signed the informed consent

Exclusion Criteria:

* Cerebral infarction, transient ischemic attack(TIA)
* Subarachnoid hemorrhage
* Proven cerebral embolism caused by tumor, Brain Trauma, cerebral parasitic disease, dysbolismus, fibrillation atrial resulted from rheumatic heart disease, coronary heart disease, and other heart diseases
* Clinical signs of infection on admission
* Pregnant or breast-feeding
* Allergic to rhubarb
* Preceding or ongoing antibiotic therapy within the last 24 h
* Participation in another interventional trial
* Immunosuppressant treatment within the last 30 days
* Combining severe clinical conditions such as liver, kidney, Hematopoietic System, endocrine system or psychological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-01

PRIMARY OUTCOMES:
The lung infection rate within 14 days after stroke onset | 14 days

SECONDARY OUTCOMES:
Global disability on modified Rankin scale at 90 days | 90 days
NIH stroke scale | 90 days
Barthel Index | 90 days
Death rate | 90 days
Syndrome score by Traditional Chinese Medicine (TCM) standard | 90 days
Changes in laboratory indexes as safety assessment, including red blood cell(RBC), white blood cell(WBC), platelet(PLT), alanine transaminase (ALT), aspartate transaminase(AST), blood urea nitrogen (BUN), creatinine(Cr) in blood samples; protein, | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Cai DF, Dai W, Chen YP, Wen M, Dai HL. [Effect and mechanism of rhubarb on fibrinolysis in secondary damaged central nerve system of rats with acute hemorrhagic stroke]. Zhongguo Zhong Xi Yi Jie He Za Zhi. 2005 Jan;25(1):38-41. Chinese. PMID 15719749